CLINICAL TRIAL: NCT00699634
Title: A Randomized Double-blind Placebo Controlled Trial Assessing the Effect of the Oral Cannabinoid Nabilone on Pain and Quality of Life in Patients With Phantom Limb Pain
Brief Title: Nabilone for the Treatment of Phantom Limb Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Valeant Canada Limited (Industry)
Responsible Party: Dr. Ryan Quinlan Skrabek, University of Manitoba
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1975; REB: B2007:129; Impact: RI07:119; Health Canada: 116697
Record Dates: First submitted 2008-06-17; First posted 2008-06-18 (Estimated); Last update posted 2011-04-29 (Estimated); Status verified 2011-04

CONDITIONS: Phantom Limb Pain; Neuropathic Pain
Keywords: Neuropathic; Pain; Phantom; Limb
MeSH Terms: conditions — Phantom Limb; Neuralgia; Pain | interventions — nabilone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Nabilone — Nabilone 0.5 mg at hs for 1 week, then 0.5 mg BID for 1 week. After a reassessment of the outcome measures, the dose is increased to 0.5 mg in the morning and 1 mg at hs for 1 week, followed by an increase to 1 mg BID in the last week of the study.
  Other Names: Cesemet

SUMMARY:
The purpose of this proposed study is to conduct a randomized double-blind placebo controlled trial assessing the benefit of nabilone in pain management and improvement of quality of life in patients with phantom limb pain.

Our Hypothesis is that the synthetic cannabinoid Nabilone will significantly reduce the phantom limb pain and improve quality of life, compared to the placebo controlled group. This will be evident by finding significant differences in Visual Analogue Scale pain scores, frequency of phantom pain episodes, the Depression, Anxiety and Stress Scale, and the Groningen Sleep Quality Scale and daily prosthetic wearing time.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed with phantom limb pain by a Rehabilitation Medicine Specialist.
* 18-70 years old.
* Any gender.
* The patient has not had resolution of their phantom limb pain with other treatments, such as a tricyclic antidepressant, or anticonvulsant medication.
* No previous use of oral cannabinoids for pain management.

Exclusion Criteria:

* The patient's pain is better explained by a treatable cause of stump pain, such as neuroma or bony overgrowth.
* Gross abnormalities on routine baseline blood work including electrolytes, urea and creatinine, a complete blood count, and liver function tests (AST ALT GGT, Alk Phos, and LDH) that are twice the limit of normal. Normal tests taken within 3 months prior to the study will be accepted if there is no history of acute illness since the time the blood was drawn.
* Heart disease. (Cannabinoids can reduce heart rate and blood pressure) Patients with heart disease will be excluded based on a history of symptomatic angina, MI or CHF as well as a clinical exam.
* Schizophrenia or other Psychotic disorder
* Severe liver dysfunction.
* History of untreated non-psychotic emotional disorders.
* Cognitive impairment.
* Major illness in another body area.
* Pregnancy.
* Nursing mothers.
* History of drug dependency.
* A known sensitivity to marijuana or other cannabinoid agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-01; Primary Completion 2011-02 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale for Pain | Baseline, 2, 4 and 6 weeks

SECONDARY OUTCOMES:
Depression Anxiety and Stress Scale | Baseline, 2, 4 and 6 weeks
Groningen Sleep Quality Scale | Baseline, 2, 4 and 6 weeks
SF-36 | Baseline, 2, 4 and 6 weeks
Frequency of phantom limb pain | Baseline, 2, 4 and 6 weeks
Daily prosthetic wearing time | Baseline, 2, 4 and 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Q Skrabek, MD, FRCPC, Principal Investigator — University of Manitoba
Locations (1):
- Rehabilitation Hospital, Winnipeg, Manitoba, Canada